CLINICAL TRIAL: NCT03857737
Title: A Study Which Compares the Long Term and Short Term Outcomes Between Endoscopic Submucosal Dissection and Surgery in the Treatment of Early Gastric Cancer
Brief Title: Endoscopic Submucosal Dissection Versus Surgery in the Treatment of Early Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Shigang Ding, Attending, Chief of the Gastrointestinal Department of Peking University Third Hospital, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUTH020301ESD
Record Dates: First submitted 2019-02-25; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Early Gastric Cancer
Keywords: early gastric cancer; endoscopic submucosal dissection; surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESD group (Experimental): This group include patients who are going to undergo endoscopic submucosal dissection for early gastric cancer.
  Interventions: Procedure: endoscopic submucosal dissection
- Surgery group (Active Comparator): This group include patients who are going to undergo surgery for early gastric cancer.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: endoscopic submucosal dissection — Endoscopic submucosal dissection is an endoscopic procedure which can achieve en bloc resection of GI tumor. ESD is characterized by three steps: injecting fluid into the submucosa to elevate the lesion from the muscle layer, circumferential cutting of the surrounding mucosa of the lesion, and subsequent dissection of the connective tissue of the submucosa beneath the lesion. The ESD procedure will be carried out by experienced endoscopists.
  Arms: ESD group
Procedure: Surgery — Surgery for EGC include Distal, proximal, or total gastrectomy, which will be performed according to the location and macroscopic tumor type by experienced surgeons.
  Arms: Surgery group

SUMMARY:
In this study, patients who are going to undergo endoscopic submucosal dissection (ESD) or surgery for early gastric cancer will be enrolled and divided into ESD group and Surgery group according to the procedure they go through. The patients will be followed up for at least 5 years after ESD or surgery. Esophagogastroduodenoscopy (EDG) and biopsy will be performed 3 months and then 6 months after ESD or surgery. Thereafter, EDG will be performed along with biopsy and abdominal computed tomography annually up to 5 years. Patients' data such as age, sex, clinical diagnosis, achievement of en-bloc resection, pathological outcomes, complications and survival condition will be prospectively collected. Statistical methods such as Student's t-test, the chi-square test, the Kaplan-Meier method and the log-rank test will be used to compare the short term and long term outcomes between the ESD group and the surgery group.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as early gastric cancer
* Willing to undergo endoscopic submucosal dissection or surgery for the treatment of early gastric cancer

Exclusion Criteria:

* Advanced stage gastric cancer
* Not willing to undergo endoscopic submucosal dissection or surgery for the treatment of early gastric cancer
* Not willing to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year OS | From March 1 2019 to December 1 2024
  5-year OS is the five year overall survival of each individual group. It will be estimated by Kaplan-Meier method, and statistical significance of differences between the two groups will be assessed using the log-rank test.
5-year DSS | From March 1 2019 to December 1 2024
  5-year DSS is the five year disease specific survival of each individual group. It will be estimated by Kaplan-Meier method, and statistical significance of differences between the two groups will be assessed using the log-rank test.

SECONDARY OUTCOMES:
Complication | From March 1 2019 to December 1 2024
  Complications were classified according to the Clavien-Dindo classification and the frequency of the complications will be compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2014 (ver. 4). Gastric Cancer. 2017 Jan;20(1):1-19. doi: 10.1007/s10120-016-0622-4. Epub 2016 Jun 24. No abstract available. PMID 27342689
- [Background] Suzuki H, Oda I, Abe S, Sekiguchi M, Nonaka S, Yoshinaga S, Saito Y, Fukagawa T, Katai H. Clinical outcomes of early gastric cancer patients after noncurative endoscopic submucosal dissection in a large consecutive patient series. Gastric Cancer. 2017 Jul;20(4):679-689. doi: 10.1007/s10120-016-0651-z. Epub 2016 Oct 8. PMID 27722825
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Pimentel-Nunes P, Dinis-Ribeiro M, Ponchon T, Repici A, Vieth M, De Ceglie A, Amato A, Berr F, Bhandari P, Bialek A, Conio M, Haringsma J, Langner C, Meisner S, Messmann H, Morino M, Neuhaus H, Piessevaux H, Rugge M, Saunders BP, Robaszkiewicz M, Seewald S, Kashin S, Dumonceau JM, Hassan C, Deprez PH. Endoscopic submucosal dissection: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2015 Sep;47(9):829-54. doi: 10.1055/s-0034-1392882. Epub 2015 Aug 28. PMID 26317585